CLINICAL TRIAL: NCT05446961
Title: Pilot Phase II Randomized, Placebo-Controlled Clinical Trial for the Prevention and Progression of SARS-CoV-2 Infection of Subjects and Patients Using a Supplement Treatment With Carnipure Tartrate ( LCLT)
Brief Title: Clinical Study to Evaluate the Effect of Food Supplement in People Infected With Coronavirus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SENAI CIMATEC (Other)
Collaborators: Hospital Espanhol (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01/2021
Record Dates: First submitted 2022-04-23; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Virus Infection
MeSH Terms: conditions — COVID-19 | interventions — Carnitine; Dosage Forms

STUDY DESIGN:
Intervention Model Description: A total of 274 subjects, will be prospectively enrolled into a pilot randomized, placebo controlled study in the two cohorts: Cohort 1: 220 healthy, SARS-CoV-2 negative, individuals (55 to 85 years old) with close contact (cohabit) to a person with newly acquired SARS-CoV-2 infection based on PCR detection and absence of antibody response; and, Cohort 2: 54 asymptomatic ( 18 to 85 years old) or symptomatic patients with mild COVID-19 that tested positive for COVID-19 by RT-PCR within the last 24 hours prior to the enrolment in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The groups will be randomized and blindly assigned to receive either the LCLT supplement (3 g per day that delivers 2 g elemental of L-carnitine) or placebo. Subjects from Cohort 2 will receive L-carnitine in addition to Standard of Care (SOC) therapy or placebo in addition tosStandard of care (SOC) therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- covid 19 LCLT supplement (Active Comparator): LCLT is made out of 68% elemental L-carnitine and 32 % Tartric acid and therefore the EFSA (European Food Safety Authority) stated that it is safety up to at least 3 g. Each 3 g of LCLT delivers 2 g of elemental L-carnitine L-carnitine and Tartric acid, 3g oral capsules daily use for 21 days
  Interventions: Dietary Supplement: LCLT : 68% elemental L-carnitine and 32 % Tartric acid
- covid 19 placebo (Placebo Comparator): The formulation will contain all salt ingredients v/v without LCLT (made out of 68% elemental L-carnitine and 32 % Tartric acid) and is replaced by Maltodextrin in the placebo capsules Placebo capsules daily for 21 days
  Interventions: Drug: Placebo
- Healthy LCLT supplement (Active Comparator): LCLT is made out of 68% elemental L-carnitine and 32 % Tartric acid and therefore the EFSA (European Food Safety Authority) stated that it is safety up to at least 3 g. Each 3 g of LCLT delivers 2 g of elemental L-carnitine L-carnitine and Tartric acid, 3g oral capsules daily use for 21 days
  Interventions: Dietary Supplement: LCLT : 68% elemental L-carnitine and 32 % Tartric acid
- Healthy Placebo (Placebo Comparator): The formulation will contain all salt ingredients v/v without LCLT (made out of 68% elemental L-carnitine and 32 % Tartric acid) and is replaced by Maltodextrin in the placebo capsules Placebo capsules daily for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: LCLT : 68% elemental L-carnitine and 32 % Tartric acid — 3 g orally capsules
  Other Names: Carnipure™ Tartrate (LCLT) formulation
  Arms: Healthy LCLT supplement; covid 19 LCLT supplement
Drug: Placebo — orally capsules
  Arms: Healthy Placebo; covid 19 placebo

SUMMARY:
The purpose of the study is to assess safety and efficacy of Carnipure tartrate (L-Carnitine and L-tartaric acid - LCLT) supplementation for SARS-Cov-2 infection

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients given written informed consent will be divided em two cohorts according to inclusion criteria.One group with patients with diagnosed mild SARS-Cov-2 infection and another with healthy contacts of patients with diagnosed mild SARS-Cov-2.

Both groups will be randomized to receive either LCLT supplementation or placebo during 21 days. After this period primary endpoints of efficacy will be assessed.

Clinical follow up evaluations will be monitored (Cohort 1 and 2), and chest tomography will be monitored in cohort 2 as well. Subjects will be followed for safety through 8 weeks (cohort 1) and 6 weeks (cohort 2) after being included into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1:

   * males and females between 55 years and 85 years of age;
   * history of close contact (cohabit) with a Family member or a person newly diagnosed with SARS-CoV-2 infection;
   * negative RT-PCR COVID-19 test on the screening immediately after contact and prior to start treatment of the study.
2. Cohort 2:

   * males and females between 18 years and 85 years of age;
   * positive RT-PCR COVID-19 test and medical history and physical exam compatible with asymptomatic or mild COVID-19 pneumonia. Evaluation of clinical outcomes: oxygen requirements, hospitalization breathless and others;
   * Female subjects of childbearing potential must :

     * have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of each study supplementation;
     * no breast-feeding;
     * agree to use one of the following methods of contraception from enrollment in study until 30 days after last supplementation (only if in sexual relationships with men): hormonal (e.g. oral, transdermal, intravaginal, implant, or injection); double barrier (i.e., condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD) or system (IUS); vasectomized partner (6 months minimum); or abstinence; bilateral tubal ligation (if no conception post-procedure); tubal occlusion; or bilateral salpingectomy. Women are considered non-child-bearing potential if they are post-menopausal (defined as at least 12 months spontaneous amenorrhea and confirmed with FSH > 40 mIU/ml) or have had documented hysterectomy and/or oophorectomy. system (IUS); vasectomized partner (6 months minimum); or abstinence; bilateral tubal ligation (if no conception post-procedure); tubal occlusion; or bilateral salpingectomy;
   * Normal laboratory values of sodium, potassium, ALT, AST, total bilirubin, alcaline phosphatase, creatinine, fasting glucose, total WBC count, hemoglobina and platelet count;
   * No medical history of alcohol or drug abuse

Exclusion Criteria:

* Hormonal replacement therapy;
* Severe COVID-19 pneumonia according to CDC criteria;
* Positive test for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies;
* Participation in another experimental protocol and/or receipt of any investigational products within the past 3 months prior to Screening;
* Immunosuppressive cytotoxic therapies (e.g., chemotherapy drugs or radiation) in the past 6 months prior to Screening;
* Subjects unable to sign the inform consent to participate into the study;
* History of any other acute or uncontrolled chronic illness (including, hypertension, cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic or renal disorders) that is not on medication regimen for at least the past 6 months;
* Medication or supplements that may interfere with the evaluation of the safety and tolerability of the study drug such as ACE Inhibitors, Angiotensin II Receptor Blockers (ARBs) (e.g. vitamin B3 and L-carnitine/acetyl-carnitine).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Number new SARS-CoV-2 cases at 21 days assessed by RT-PCR | 21 days
  Number new SARS-CoV-2 cases at 21 days assessed by RT-PCR
Number of participants with severe COVID pneumonia measured by the presence of ground-glass opacity, consolidations, parenchymal bands, and crazy-paving pattern in chest tomography | 21 days
  Number of participants with severe COVID pneumonia measured by the presence of ground-glass opacity, consolidations, parenchymal bands, and crazy-paving pattern in chest tomography

SECONDARY OUTCOMES:
Levels of C-Reactive Protein (CRP) from baseline to 7, 14 and 21 days | 1,7,14 and 21 days
  Levels of C-Reactive Protein (CRP) from baseline to 7, 14 and 21 days
Total white blood count (1000 per mm³) from baseline to 7, 14 and 21 days | 1,7,14 and 21 days
  Total white blood count (1000 per mm³) from baseline to 7, 14 and 21 days
Levels of plasma ACE1 and ACE2 receptors from baseline to 7, 14 and 21 days | 1, 7, 14 and 21 days
  Levels of plasma ACE1 and ACE2 receptors from baseline to 7, 14 and 21 days
ACE1/ACE2 ratio from baseline to 7, 14 and 21 days days until the end of the study of each cohort | 1, 7, 14 and 21 days
  ACE1/ACE2 ratio from baseline to 7, 14 and 21 days days until the end of the study of each cohort
ACE1, ACE2, TMPRSS2 and furin gene expression levels from baseline to 21 days placebo in each cohort | 1 and 21 days
  ACE1, ACE2, TMPRSS2 and furin gene expression levels from baseline to 21 days
Presence of presence of ground-glass opacity, consolidations, parenchymal bands, and crazy-paving pattern in chest tomography from baseline to 7, 14 and 21 days | 1, 7, 14 and 21 days
  Presence of presence of ground-glass opacity, consolidations, parenchymal bands, and crazy-paving pattern in chest tomography from baseline to 7, 14 and 21 days
Levels of inflammatory cytokines IL-6, IL-2, IL-7, IL-10,granulocyte-colony stimulating factor (GM-CSF), interferon-γ (IFN-γ) and Tumor Necrosis Factor (TNF-α) from baseline to 7, 14 and 21 days | 1,7,14 and 21 days
  Levels of inflammatory cytokines IL-6, IL-2, IL-7, IL-10,granulocyte-colony stimulating factor (GM-CSF), interferon-γ (IFN-γ) and Tumor Necrosis Factor (TNF-α) from baseline to 7, 14 and 21 days
Levels of total white blood count (1000 per mm³) from baseline to 7, 14 and 21 days Days 1, 7, 14 and 21 days after the administration of supplement or placebo in each cohort | 1,7,14 and 21 days
  Levels of total white blood count (1000 per mm³) from baseline to 7, 14 and 21 days
Levels of hemoglobin count (g/dl) from baseline to 7, 14 and 21 days Days 1, 7, 14 and 21 days after the administration of supplement or placebo in each cohort | 1,7,14 and 21 days
  Levels of hemoglobin count (g/dl) from baseline to 7, 14 and 21 days
Total platelets count (1000 per mm³) from baseline to 7, 14 and 21 days Days 1, 7, 14 and 21 days after the administration of supplement or placebo in each cohort | 1,7,14 and 21 days
  Total platelets count (1000 per mm³) from baseline to 7, 14 and 21 days
Levels of fibrinogen (g/L) from baseline to 7, 14 and 21 days Days 1, 7, 14 and 21 days after the administration of supplement or placebo in | 1,7,14 and 21 days
  Levels of fibrinogen (g/L) from baseline to 7, 14 and 21 days
Levels of D-Dimer (µg/mL) from baseline to 7, 14 and 21 days | 1,7,14 and 21 days
  Levels of D-Dimer (µg/mL) from baseline to 7, 14 and 21 days
Levels of Ferritin (µg/mL) from baseline to 7, 14 and 21 days Days 1, 7, 14 and 21 days after the administration of supplement or placebo in each cohort | 1,7,14 and 21 days
  Levels of Ferritin (µg/mL) from baseline to 7, 14 and 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Badaró, Ph.D, Principal Investigator — SENAI CIMATEC
Locations (1):
- Senai Cimatec, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] FRITZ IB. Action of carnitine on long chain fatty acid oxidation by liver. Am J Physiol. 1959 Aug;197:297-304. doi: 10.1152/ajplegacy.1959.197.2.297. No abstract available. PMID 13825279
- [Background] Brass EP. Pharmacokinetic considerations for the therapeutic use of carnitine in hemodialysis patients. Clin Ther. 1995 Mar-Apr;17(2):176-85; discussion 175. doi: 10.1016/0149-2918(95)80017-4. PMID 7614519
- [Background] Kraemer WJ, Volek JS, Dunn-Lewis C. L-carnitine supplementation: influence upon physiological function. Curr Sports Med Rep. 2008 Jul-Aug;7(4):218-23. doi: 10.1249/JSR.0b013e318180735c. PMID 18607224
- [Background] Ozturk MA, Kardas Z, Kardas F, Gunes T, Kurtoglu S. Effects of L-carnitine supplementation on respiratory distress syndrome development and prognosis in premature infants: A single blind randomized controlled trial. Exp Ther Med. 2016 Mar;11(3):1123-1127. doi: 10.3892/etm.2015.2964. Epub 2015 Dec 29. PMID 26998047
- [Result] Verity R, Okell LC, Dorigatti I, Winskill P, Whittaker C, Imai N, Cuomo-Dannenburg G, Thompson H, Walker PGT, Fu H, Dighe A, Griffin JT, Baguelin M, Bhatia S, Boonyasiri A, Cori A, Cucunuba Z, FitzJohn R, Gaythorpe K, Green W, Hamlet A, Hinsley W, Laydon D, Nedjati-Gilani G, Riley S, van Elsland S, Volz E, Wang H, Wang Y, Xi X, Donnelly CA, Ghani AC, Ferguson NM. Estimates of the severity of coronavirus disease 2019: a model-based analysis. Lancet Infect Dis. 2020 Jun;20(6):669-677. doi: 10.1016/S1473-3099(20)30243-7. Epub 2020 Mar 30. PMID 32240634
- [Result] Hamming I, Timens W, Bulthuis ML, Lely AT, Navis G, van Goor H. Tissue distribution of ACE2 protein, the functional receptor for SARS coronavirus. A first step in understanding SARS pathogenesis. J Pathol. 2004 Jun;203(2):631-7. doi: 10.1002/path.1570. PMID 15141377
- [Result] Ciaglia E, Vecchione C, Puca AA. COVID-19 Infection and Circulating ACE2 Levels: Protective Role in Women and Children. Front Pediatr. 2020 Apr 23;8:206. doi: 10.3389/fped.2020.00206. eCollection 2020. No abstract available. PMID 32391299